CLINICAL TRIAL: NCT07262307
Title: Evaluation of PEEK Versus Titanium Bar Attachments With Implant Assisted Mandibular Complete Overdenture Fabricated by CAD/CAM Technology
Acronym: Evaluation
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Nour Elhouda, Assistant lecturer, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2140
Record Dates: First submitted 2025-09-07; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-02

CONDITIONS: Edentulism in Lower Jaw

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Evaluation of PEEK material (Experimental): digital fabrications techniques
  Interventions: Device: implant overdenture
- Group Ӏ (control group): Six patients will receive digital mandibular implant overdenture assisted b (Active Comparator): • Clinical evaluation
  Interventions: Device: implant overdenture
- PEEK group new material (Experimental)
  Interventions: Device: implant overdenture
- PEEK material study group (Experimental)
  Interventions: Device: implant overdenture

INTERVENTIONS:
Device: implant overdenture — using of CAD/CAM with new material and digital fabrication techniques

SUMMARY:
Evaluation of PEEK versus Titanium Bar Attachments with Implant Assisted Mandibular Complete Overdenture fabricated by CAD/CAM Technology measuring retention of the overdenture and implant evaluation for 6 months and one year

ELIGIBILITY:
Inclusion Criteria:

* • Completely edentulous patients free from systemic diseases that may affect soft or hard tissue healing.

  * Patient's age ranges from 40 to 60 years old.
  * The bone quality and quantity of the mandibular alveolar ridge must fulfill the criteria for implant placement.
  * They have normal class Ӏ maxilla-mandibular relationship and sufficient inter-arch space with at least 25mm for bar attachment.
  * They have good oral hygiene.

Exclusion Criteria:

* Systemic disorders that may influence soft or hard tissue healing as oral diseases.
* Patients with history of radiation therapy in the head and neck region.
* Patients with neurological or psychological problems that may impair good oral hygiene.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
retention of mandibular overdenture | 6 months and 12 months post-insertion
  Retention of the mandibular implant-assisted complete overdenture will be measured using a digital force meter. Measurements will be taken at 6 months and 12 months after denture insertion.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Tanta, Elgharbiy, Egypt

DOCUMENTS (7):
  • Study Protocol: Evaluation of digitalPEEK Versus Titanium Bar Attachments (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_000.pdf
  • Study Protocol: . Evaluation of digitalPEEK Versus Titanium Bar Attachments (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_001.pdf
  • Study Protocol and Statistical Analysis Plan: Evaluation of PEEK Versus Titanium Bar Attach (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_SAP_002.pdf
  • Study Protocol: Evaluation of digital PEEK Versus Titanium Bar Attachments (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_003.pdf
  • Study Protocol: Evaluation of digital PEE Versus Titanium Bar Attachments (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_004.pdf
  • Study Protocol and Statistical Analysis Plan: . Evaluation of Digit PEEK Versus Titanium Bar Attachments (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_SAP_005.pdf
  • Study Protocol: . Evaluation of digital PEE Versus Titanium Bar Attachments (2024-02-20): https://cdn.clinicaltrials.gov/large-docs/07/NCT07262307/Prot_006.pdf